CLINICAL TRIAL: NCT01330966
Title: A Phase II Study of Pazopanib in the Treatment of Surgically Unresectable or Metastatic Chondrosarcoma
Brief Title: Study of Pazopanib in the Treatment of Surgically Unresectable or Metastatic Chondrosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emerald Clinical Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAPSMCS1002
Record Dates: First submitted 2011-04-06; First posted 2011-04-07 (Estimated); Results first posted 2020-02-12 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Chondrosarcoma; Metastatic Chondrosarcoma
Keywords: surgically unresectable chondrosarcoma
MeSH Terms: conditions — Chondrosarcoma | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pazopanib (Experimental): Pazopanib 800 mg orally once daily will be started on Cycle 1 Day 1 and will be administered continuously for a 28-day cycle.
  Interventions: Drug: pazopanib

INTERVENTIONS:
Drug: pazopanib — Pazopanib 800 mg orally once daily will be started on Cycle 1 Day 1 and will be administered continuously for a 28-day cycle.
  Other Names: Votrient

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of single agent pazopanib in subjects with chondrosarcoma.

DETAILED DESCRIPTION:
This research study is being conducted in adult subjects with a type of bone cancer called chondrosarcoma that has spread to other parts of the body and is not able to be removed with surgery. There is only one study drug that will be used in this study. It is a drug that interferes with cell communication and growth, taken orally. The study drug is called pazopanib.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age > or = to 18 years.
* Histologically confirmed diagnosis of conventional chondrosarcoma of any grade.
* Surgically unresectable or metastatic disease.
* Any number of prior treatment regimens, including treatment naive subjects. Prior treatment with tyrosine kinase inhibitors is permitted.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Measurable or evaluable (non-measurable) disease per RECIST guidelines version 1.1.
* Adequate organ system function determined within 14 days prior to first dose of study treatment.
* Left ventricular ejection fraction > 50% or the institutional LLN within 28 days prior to the first dose of study treatment.
* Females must either be of non-child bearing potential or have a negative serum pregnancy test within 7 days prior to the first dose of study treatment.

Exclusion Criteria:

* Prior treatment with pazopanib.
* Mesenchymal, dedifferentiated, and extraskeletal myxoid chondrosarcoma subtypes.
* Prior malignancy (Note: subjects who have had another malignancy and have been disease-free for 3 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible).
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, unless previously treated, asymptomatic, and off steroids and anti-seizure medication for 6 months prior to first dose of study drug.
* Clinically significant gastrointestinal (GI) abnormalities that may increase the risk for GI bleeding.
* Clinically significant GI abnormalities that may affect absorption of investigational product.
* Presence of uncontrolled infection.
* Corrected QT interval > 480 msecs using Bazett's formula.
* History of certain cardiovascular conditions within the past 6 months.
* Poorly controlled hypertension [defined as systolic blood pressure of > or = 140 mmHg or diastolic blood pressure of > or = 90 mmHg].
* History of cerebrovascular accident including transient ischemic attack, pulmonary embolism, or untreated deep venous thrombosis within the past 6 months.
* Prior major surgery or trauma within 28 days prior to the first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer.
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage.
* Hemoptysis in excess of 2.5 mL within 8 weeks of first dose of study drug.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Unable or unwilling to discontinue use of prohibited medications for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of study treatment.
* Radiation therapy, surgery (except major surgery), tumor embolization, chemotherapy, immunotherapy, biologic therapy, investigational therapy, or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug.
* Any ongoing toxicity from prior anti-cancer therapy that is > Grade 1 and/or that is progressing in severity, except alopecia.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to pazopanib or excipients that contraindicates participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-04; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Staddon, MD, Study Chair — Pennsylvania Oncology Hematology Associates; Warren Chow, MD, Study Chair — City of Hope Medical Center
Locations (7):
- United States (6):
  - City of Hope, Duarte, California
  - Edward Cancer Center, Naperville, Illinois
  - University of Iowa, Iowa City, Iowa
  - Mayo Clinic, Rochester, Minnesota
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - MD Anderson, Houston, Texas
- University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital, Queen Elizabeth Medical Centre, Edgbaston, Birmingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Pazopanib: Pazopanib 800 mg orally once daily will be started on Cycle 1 Day 1 and will be administered continuously for a 28-day cycle. Study treatment may continue until disease progression or unacceptable toxicity.
  pazopanib: Pazopanib 800 mg orally once daily will be started on Cycle 1 Day 1 and will be administered continuously for a 28-day cycle.
Period: Overall Study
Arm/Group | Pazopanib
Started | 47
Completed | 42 (Tumor responses evaluable in 42 of 47 pts; 5 pts discontinued prior to first tumor assessment.)
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Pazopanib
Number analyzed (Participants) | 47
Age, Continuous [Median (Full Range); unit: years] | 58 [32 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 39
  Asian | 2
  Black or African American | 3
  Hispanic | 3
Region of Enrollment [Number; unit: participants]
  United States | 45
  United Kingdom | 2

OUTCOME MEASURES:

1. Primary Outcome: Disease Control at Week 16
Description: Disease control at week 16 defined as complete response (CR), Disappearance of all target lesions; plus partial response (PR), At least a 30% decrease in the sum of diameters of the target lesions taking as reference the Baseline sum diameters; plus stable disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum diameters while on the study; where tumor response is defined by RECIST (Response Evaluation Criteria in Solid Tumors) guidelines version 1.1. Repeat radiologic imaging is performed after every 2 cycles of treatment (approximately every 8 weeks).
Time Frame: Assessed at week 16 of study treatment
Population: Tumor responses were evaluable in 42 out of 47 patients; 5 patients discontinued prior to the first tumor assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of CR+PR+SD
Arm/Group | Pazopanib
Number analyzed (Participants) | 42
Percentage of CR+PR+SD | 43 [28 to 58]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: The time origin for PFS will be cycle 1 day 1. Repeat radiologic imaging will be conducted after every 2 cycles of treatment (approximately every 8 weeks). No upper limits of duration of assessment are identified or defined in the protocol.
Time Frame: Cycle 1 day 1 until the subject experiences disease progression
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib
Number analyzed (Participants) | 47
months | 7.9 [3.7 to 12.6]

3. Secondary Outcome: Overall Survival (OS)
Description: The time origin for OS will be cycle 1 day 1. Subjects will be followed until 6 months after end of treatment, lost to follow-up, or withdrawal of consent. No upper limits of duration of assessment are identified or defined in the protocol.
Time Frame: Cycle 1 day 1 until 6 months after end of treatment, is lost to follow-up, or withdraws consent
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib
Number analyzed (Participants) | 47
months | 17.6 [11.3 to 35.0]

ADVERSE EVENTS:
Time Frame: For each subject, adverse events were collected beginning at the start of study treatment until 30 days after discontinuation of treatment.
Arm/Group | Pazopanib
All-Cause Mortality (participants affected / at risk) | 1/47
Serious Adverse Events (participants affected / at risk) | 19/47
Other Adverse Events (participants affected / at risk) | 39/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pazopanib (N=47)
Abdominal abscess (Infections and infestations) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine amino transferase increased (Investigations) | 1 (2)
Anorectal infection (Infections and infestations) | 1 (1)
Central nervous system hemorrhage (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Embolism (Vascular disorders) | 3 (4)
Gastronomy tube site reaction (Injury, poisoning and procedural complications) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperbilirubin (Hepatobiliary disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Troponin increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pazopanib (N=47)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 4 (4)
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 11 (13)
Diarrhoea (Gastrointestinal disorders) | 22 (43)
Dyspepsia (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 24 (35)
Oral dysaesthesia (Gastrointestinal disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 3 (5)
Vomiting (Gastrointestinal disorders) | 10 (14)
Fatigue (General disorders) | 21 (31) — Fatigue
Oedema peripheral (General disorders) | 8 (11)
Bronchitis (Infections and infestations) | 2 (2)
Gingivitis (Infections and infestations) | 2 (2)
Mucosal infection (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (5)
Contusion (Injury, poisoning and procedural complications) | 4 (4)
Aspatartate amino transferase increased (Investigations) | 6 (7)
Blood bilirubin increased (Investigations) | 3 (4)
Neutrophil count decreased (Investigations) | 5 (9)
Platelet count decreased (Investigations) | 5 (10)
Weight decreased (Investigations) | 14 (19)
White blood cell count decreased (Investigations) | 3 (8)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Hypoabluminanemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (13)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 8 (9)
Headache (Nervous system disorders) | 6 (6)
Neuralgia (Nervous system disorders) | 2 (3)
Haematuria (Renal and urinary disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hair colour changes (Skin and subcutaneous tissue disorders) | 10 (10)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (4)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT01330966/Prot_SAP_000.pdf